CLINICAL TRIAL: NCT03729596
Title: A Phase 1/2, First-in-Human, Open-Label, Dose-Escalation Study of MGC018 (Anti-B7-H3 Antibody Drug Conjugate) Alone and in Combination With MGA012 (Anti-PD-1 Antibody) in Patients With Advanced Solid Tumors
Brief Title: MGC018 With or Without MGA012 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGC018-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-02 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Cancer; Melanoma; Advanced Solid Tumor, Adult; Metastatic Castrate Resistant Prostate Cancer; Non Small Cell Lung Cancer
Keywords: antibody-drug conjugate (ADC); B7-H3
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Dose escalation will use a 3+3+3 design to identify an MAD or MTD, followed by a Cohort Expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1 (Experimental): 0.5 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- Cohort 2 (Experimental): 1.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- Cohort 3 (Experimental): 2.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- Cohort 4 (Experimental): 3.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- Cohort 5 (Experimental): 4.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- mCRPC expansion (Experimental): 3.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- NSCLC expansion (Experimental): 3.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- TNBC expansion (Experimental): 3.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- Melanoma expansion (Experimental): 3.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine
- SCCHN expansion (Experimental): 3.0 mg/kg IV every 3 weeks
  Interventions: Biological: vobramitamab duocarmazine

INTERVENTIONS:
Biological: vobramitamab duocarmazine — Anti-B7H3 antibody drug conjugate
  Other Names: MGC018

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics (PK) pharmacodynamics and preliminary antitumor activity of vobramitamab duocarmazine (MGC018) in patients with advanced solid tumors. Patients with solid tumors will be enrolled in the Dose Escalation Phase; Cohort Expansion will include metastatic castrate-resistant prostate cancer (mCRPC), non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC), squamous cell carcinoma of the head and neck (SCCHN), and melanoma. Patients who do not experience unacceptable toxicity or meet criteria for permanent discontinuation may undergo additional cycles for up to two years. Patients in Cohort Expansion will be followed for survival every 3 months for 2 years following last dose.

ELIGIBILITY:
Inclusion Criteria:

* Tissue specimen available for retrospective analysis of B7-H3 and PD-L1 expression.
* Eastern Cooperative Oncology Group performance status of ≤2
* Life expectancy ≥ 12 weeks for dose escalation phase and ≥ 24 weeks for cohort expansion phase
* Measurable disease. Prostate cancer patients with bone only disease are eligible.
* Acceptable laboratory parameters and adequate organ reserve.
* Dose Escalation Phase: Patients with histologically proven, unresectable, locally advanced or metastatic solid tumors for whom no therapy with demonstrated clinical benefit is available.

Module A Cohort Expansion:

* mCRPC that has progressed with one prior line of chemotherapy for metastatic disease and no more than two prior lines of anti-hormonal therapy.
* NSCLC: metastatic disease after standard cytotoxic, targeted, and biologic or checkpoint inhibitor therapy. No more than 2 prior lines of chemotherapy.
* TNBC: Locally advance or metastatic disease that has progressed following at least one systemic therapy.
* SCCHN that has progressed during or following at least one systemic therapy for metastatic or recurrent unresectable disease. No more than 2 prior lines of chemotherapy.
* Melanoma that has progressed during or following at least one systemic treatment for unresectable locally advanced or metastatic disease. Patients who are intolerant of or refused standard therapy are eligible.

Exclusion Criteria:

* Patients with history of prior central nervous system (CNS) metastasis must have been treated, be asymptomatic, and not have concurrent treatment for CNS disease, progression of CNS metastases on MRI, CT or PET within 6 months, or history of leptomeningeal disease or cord compression at the time of enrollment.
* Prior treatment with B7-H3 targeted agents for cancer.
* Treatment with systemic cancer therapy, biologic agents, or anti-hormonal therapy (mCRPC) within 4 weeks, prior small molecule targeted or kinase inhibitors within 14 days or 5 half-lives, prior radioligand within 6 months
* Clinically significant cardiovascular disease.
* Clinically significant pulmonary compromise or requirement for supplemental oxygen.
* History of clinically-significant cardiovascular disease, including but not limited to pericarditis or pericardial effusion.
* Active viral (including confirmed or presumed COVID-19), bacterial, or systemic fungal infection requiring parenteral treatment within 7 days of first study drug administration.
* Known history of hepatitis B or C infection or known positive test for hepatitis B surface antigen or core antigen, or hepatitis C polymerase chain reaction.
* Known positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome.
* Major trauma or major surgery within 4 weeks of first study drug administration.
* Clinically significant venous insufficiency.
* > Grade 1 peripheral neuropathy.
* Evidence of pleural effusion.
* Evidence of ascites.
* Serum testosterone >50 ng/dl or >1.7 nmol/L in mCRPC in Module A Cohort Expansion Phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ward, M.D., Study Director — MacroGenics
Locations (21):
- United States (9):
  - UCLA Department of Medicine - Hematology/Oncology, Santa Monica, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - START Midwest, Grand Rapids, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialist, Fairfax, Virginia
- Australia (4):
  - St Vincent's Health Network (Kinghorn Cancer Centre), Darlinghurst
  - Austin Health - Olivia Newton John Cancer Center, Heidelberg
  - Calvary Mater NewCastle, Waratah
  - The University of Queensland - Princess Alexandra Hospital (PAH), Woolloongabba
- Poland (4):
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie Oddział Kliniczny Onkologii, Krakow
  - Med-Polonia Sp. z o.o., Poznan
  - Magodent Sp. z o.o. Szpital Elbląska Oddział Onkologii Klinicznej/ Chemioterapii, Warsaw
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy Oddział Badań Wczesnych Faz, Warsaw
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Català D'Oncologia - Hospital Universitari Germans Trias I Pujol, Barcelona
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Ruber Internacional, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Module B of the study was never initiated. There were no participants enrolled.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
Started | 3 | 6 | 7 | 7 | 6 | 41 | 21 | 18 | 21 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 7 | 7 | 6 | 41 | 21 | 18 | 21 | 13
Not completed — Death | 3 | 5 | 4 | 1 | 0 | 34 | 18 | 14 | 19 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — protocol amendment | 0 | 1 | 3 | 6 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 2 | 3
Not completed — study terminated by sponsor | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion | Total
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 6 | 41 | 21 | 18 | 21 | 13 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.42) | 56.5 (11.98) | 64.0 (11.72) | 63.0 (10.47) | 65.5 (8.09) | 69.6 (6.97) | 60.7 (8.13) | 49.0 (12.58) | 64.0 (15.09) | 63.2 (10.35) | 62.9 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 1 | 1 | 0 | 12 | 18 | 5 | 4 | 48
  Male | 2 | 2 | 5 | 6 | 5 | 41 | 9 | 0 | 16 | 9 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 3 | 2 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 12
  Asian | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 5
  White | 3 | 3 | 5 | 4 | 4 | 37 | 19 | 15 | 19 | 12 | 121
  Other | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 7 | 7 | 6 | 21 | 2 | 2 | 6 | 0 | 60
  Poland | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 1 | 1 | 26
  Australia | 0 | 0 | 0 | 0 | 0 | 11 | 6 | 5 | 10 | 3 | 35
  Spain | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 4 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events of Vobramitamab Duocarmazine as Assessed by CTCAE v4.03
Description: Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit.
Time Frame: Throughout the study up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 6 | 41 | 21 | 18 | 21 | 13
Participants | 3 | 6 | 7 | 7 | 6 | 41 | 21 | 18 | 21 | 13

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: Number of participants with severe side effects from study treatment during the DLT evaluation period (6 weels)
Time Frame: up to 42 days from first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 6
Participants | 0 | 1 | 1 | 0 | 1

3. Secondary Outcome: Best Overall Response (BOR) of Vobramitamab Duocarmazine
Description: The best response recorded from the start of the study treatment until the end of treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1, taking into account any requirement for confirmation of response.
  Complete response (CR) is defined as disappearance of all target and non-target lesions.
  Partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, no progression of non-target lesions, and no new lesions.
  Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or unequivocal progression of non-target lesions, or appearance of new lesions.
  Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify as progression.
  Not evaluable (NE) is where the response cannot be determined.
Time Frame: Throughout the study for up to 24 months
Population: All participants who received at least one dose of study drug, had baseline measurable or non-measurable disease, and had at least one post-baseline radiographic tumor assessment or discontinued treatment due to clinical progressive disease or death.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 5 | 41 | 20 | 16 | 21 | 13
Participants
  Partial Response | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 1 | 1
  Stable Disease | 2 | 3 | 3 | 4 | 3 | 28 | 8 | 8 | 12 | 7
  Progressive Disease | 1 | 3 | 0 | 2 | 1 | 11 | 7 | 8 | 8 | 3
  Not Evaluated | 0 | 0 | 4 | 1 | 0 | 0 | 2 | 0 | 0 | 2

4. Secondary Outcome: Objective Response Rate (ORR) of Vobramitamab Duocarmazine
Description: The percentage of participants who achieve a complete response (CR or partial response (PR) to treatment with vobramitamab duocarmazine
Time Frame: Efficacy evaluations every 9 weeks throughout the study for up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 6 | 41 | 21 | 18 | 21 | 13
percentage of participants | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 41.0] | 0 [0 to 41.0] | 20 [0.5 to 71.6] | 4.9 [0.6 to 16.5] | 15.0 [3.2 to 37.9] | 0 [0 to 20.6] | 4.8 [0.1 to 23.8] | 7.7 [0.2 to 36.0]

5. Secondary Outcome: Progression Free Survival (PFS) of Vobramitamab Duocarmazine
Description: PFS is calculated from the first dose date until the date of first documented PD using RECIST v1.1, or death from any cause, whichever occurs first.
  Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or unequivocal progression of non-target lesions, or appearance of new lesions. Median PFS and 95% CI is estimated using the Kaplan-Meier method.
Time Frame: Every 9 weeks for up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
Number analyzed (Participants) | 3 | 5 | 2 | 3 | 2 | 29 | 15 | 18 | 17 | 10
months | 2.8 [1.28 to 3.45] | 2.0 [0.76 to NA] — upper bound could not be calculated due to lack of survival events | 4.0 [0.85 to NA] — upper bound could not be calculated due to lack of survival events | 6.3 [1.38 to 6.31] | 4.0 [1.41 to NA] — upper bound could not be calculated due to lack of survival events | 5.5 [2.92 to 8.28] | 4.0 [2.10 to 4.17] | 2.4 [2.04 to 4.17] | 3.5 [2.00 to 7.33] | 3.3 [1.02 to 4.17]

6. Secondary Outcome: Median Duration of Response (DoR) of Vobramitamab Duocarmazine
Description: Median DoR assessed as the time from the date of initial objective response to the date of first documented PD, per RECIST v1.1, or the date of death from any cause, whichever occurs first.
  Median DoR and 95% CI is estimated using the Kaplan-Meier method.
Time Frame: Throughout the study for up to 48 months
Population: Participants who experienced a complete or partial response to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 1 | 1
months |  |  |  |  | 5.32 [NA to NA] — Data reported for a single participant. | 5.3 [4.27 to 6.28] | NA [4.53 to NA] — The upper bound of the CI could not be estimated due to insufficient number of participants with events |  | 10.28 [NA to NA] — Data reported for a single participant. | 2.10 [NA to NA] — Data reported for a single participant.

7. Secondary Outcome: Median Overall Survival (OS) of Vobramitamab Duocarmazine
Description: Median OS assessed as the time from the first dose date to the date of death from any cause, using the Kaplan-Meier method for estimating median and confidence interval. .
Time Frame: Every 9 weeks for up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
Number analyzed (Participants) | 3 | 6 | 7 | 7 | 6 | 41 | 21 | 18 | 21 | 13
months | 3.5 [2.83 to 11.24] | 5.7 [2.14 to NA] — Could not be estimated due to insufficient number of participants with events | 13.1 [0.85 to 13.14] | NA [8.48 to NA] — Could not be estimated due to insufficient number of participants with events | NA [NA to NA] — Could not be estimated due to insufficient number of participants with events | 12.3 [5.52 to 14.55] | 7.0 [4.01 to 8.44] | 5.8 [3.32 to 15.51] | 9.4 [5.78 to 10.74] | 5.1 [1.05 to NA] — Could not be estimated due to insufficient number of participants with events

8. Secondary Outcome: PSA Response Rate
Description: Percent of prostate cancer patients with at least 50% reduction in prostate-specific antigen (PSA) with confirmation at least 3 weeks later
Time Frame: Every 3 weeks up to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- mCRPC: Participants in cohort expansion with metastatic castration-resistant prostate cancer.
Arm/Group | mCRPC
Number analyzed (Participants) | 41
Participants | 18

9. Secondary Outcome: Best PSA Response
Description: For prostate cancer patients, the greatest change from baseline in PSA.
Time Frame: Every 3 weeks up to 24 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | mCRPC
Number analyzed (Participants) | 41
ng/mL | -43.7 (44.43)

10. Secondary Outcome: Mean Area Under the Curve (AUC) of Vobramitamab Duocarmazine Antibody Drug Conjugate (ADC)
Description: Area under the plasma concentration versus time curve of vobramitamab duocarmazine
Time Frame: At baseline, Cycle 1, Day 1: 1 hour, 4 hours after the first dose, Day 2, Day 3, Day 7, Day 14 and Cycle 2 Day 1 (approximately 21 days after the first dose).
Population: All participants who received at least one dose of study treatment, date and time of dose administration and relative PK sample collection are known and have sufficient concentration data to derive the PK parameter. One participant assigned to Cohort 4 (3.0 mg/kg dose) was actually treated at the Cohort 3 dose of 2.0 mg/kg and is therefore included in Cohort 3 for the purposes of this analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL*day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 8 | 120 | 6
mcg/mL*day | 10.6 (6.54) | 51.5 (19.2) | 119 (48.7) | 140 (34.9) | 227 (105)

11. Secondary Outcome: Mean AUC of Duocarmycin
Description: Area under the plasma concentration versus time curve of duocarmycin (unconjugated payload) in the bloodstream
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL*day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 8 | 120 | 6
ng/mL*day | 0.0448 (0.023) | 0.101 (0.0668) | 0.0512 (0.0454) | 0.657 (0.0349) | 0.0268 (0.031)

12. Secondary Outcome: Mean Maximum Concentration Vobramitamab Duocarmazine ADC
Description: Maximum Plasma Concentration of vobramitamab duocarmazine ADC in the bloodstream
Time Frame: At baseline, Cycle 1, Day 1, 1 and 4 hours after the end of infusion, Day 2, and Day 3.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 8 | 120 | 6
mcg/mL | 7.69 (1.98) | 23.4 (4.08) | 43.4 (14) | 59 (11) | 76.6 (22.4)

13. Secondary Outcome: Mean Maximum Concentration Duocarmycin
Description: Maximum Plasma Concentration of vobramitamab duocarmazine ADC in the bloodstream
Time Frame: At baseline, Cycle 1, Day 1, 1 and 4 hours after the end of infusion, Day 2, and Day 3.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 8 | 120 | 6
ng/mL | 0.0243 (0.0225) | 0.0274 (0.016) | 0.0512 (0.0454) | 0.657 (0.0349) | 0.0571 (0.00757)

14. Secondary Outcome: Mean Trough Concentration of Vobramitamab Duocarmazine ADC
Description: Average trough plasma concentration of vobramitamab duocarmazine ADC in the bloodstream.
Time Frame: At baseline, and before subsequent infusion Cycle 2, Day 1 (Study Day 22).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 8 | 120 | 6
mcg/mL | 0.00928 (0.0129) | 0.0415 (0.0415) | 0.123 (0.652) | 0.157 (0.119) | 0.313 (0.323)

15. Secondary Outcome: Mean Trough Concentration of Duocarmycin
Description: Average trough plasma concentration of duocarmycin unconjugated payload in the bloodstream.
Time Frame: At baseline, and before subsequent infusion Cycle 2, Day 1 (Study Day 22).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 8 | 120 | 6
ng/mL | 0.000243 (0.000107) | 0.00074 (0.000532) | 0.00226 (0.00244) | 0.00185 (0.000658) | 0.00194 (0.000973)

16. Secondary Outcome: Number of Participants Who Develop MGC018 Anti-drug Antibodies
Description: Shifts in MGC018 anti-drug antibodies after treatment with vobramitamab duocarmazine
Time Frame: Every 3 weeks through end of treatment, up to 24 months
Population: All participants who received at least one dose of study treatment and have at least one ADA sample sufficient for analysis. There were 3 missing samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 7 | 118 | 6
Participants
  Negative at baseline, negative post baseline | 2 | 5 | 6 | 102 | 6
  Negative at baseline, positive post baseline | 1 | 1 | 0 | 12 | 0
  missing post baseline data | 0 | 0 | 1 | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the time of first dose through 28 days after the last dose of study treatment or until the start of another anti-cancer treatment, up to 25 months. All cause mortality was assessed from the time of first dose until death, or participant withdrawal of consent, or the end of the study, whichever was earlier, up to 25 months.
Description: Adverse events are based on physical findings, patient reports, and significant laboratory values.
  Progression of neoplasm causing hospitalization or death is an antitumor activity outcome and not an SAE, unless considered drug-related by the investigator.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | mCRPC Expansion | NSCLC Expansion | TNBC Expansion | Melanoma Expansion | SCCHN Expansion
All-Cause Mortality (participants affected / at risk) | 3/3 | 5/6 | 4/7 | 1/7 | 0/6 | 34/41 | 18/21 | 14/18 | 19/21 | 9/13
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/6 | 3/7 | 2/7 | 2/6 | 23/41 | 10/21 | 6/18 | 6/21 | 5/13
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7 | 7/7 | 6/6 | 41/41 | 21/21 | 18/18 | 21/21 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=7) | Cohort 4 (N=7) | Cohort 5 (N=6) | mCRPC Expansion (N=41) | NSCLC Expansion (N=21) | TNBC Expansion (N=18) | Melanoma Expansion (N=21) | SCCHN Expansion (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis pasteurella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=7) | Cohort 4 (N=7) | Cohort 5 (N=6) | mCRPC Expansion (N=41) | NSCLC Expansion (N=21) | TNBC Expansion (N=18) | Melanoma Expansion (N=21) | SCCHN Expansion (N=13)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3 | 3 | 20 | 8 | 7 | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 4 | 2 | 12 | 2 | 8 | 5 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 3 | 4 | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 5 | 1 | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 6 | 2 | 1 | 3 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 5 | 1 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 2 | 3 | 15 | 7 | 3 | 9 | 6
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 9 | 3 | 2 | 3 | 4
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 0 | 7 | 2 | 2 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3 | 10 | 3 | 0 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 5 | 4 | 2 | 4 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 2 | 5 | 3 | 23 | 14 | 6 | 9 | 4
Oedema peripheral (General disorders) | 0 | 1 | 1 | 3 | 0 | 14 | 5 | 5 | 7 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 4 | 3 | 2 | 6
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 4 | 6 | 1 | 3 | 2 | 0
Chills (General disorders) | 1 | 1 | 2 | 0 | 2 | 3 | 1 | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 4 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 2 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 5 | 2 | 7 | 0 | 1 | 4 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 3 | 0 | 9 | 1 | 3 | 8 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 2 | 1 | 10 | 5 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 2 | 1 | 0 | 9 | 1 | 2 | 4 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 2 | 1 | 7 | 1 | 1 | 3 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 9 | 1 | 2 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 6 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 1 | 14 | 7 | 7 | 5 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 4 | 2 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 16 | 3 | 3 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 18 | 4 | 2 | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 9 | 2 | 5 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 4 | 5 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 4 | 2 | 19 | 9 | 5 | 11 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 3 | 2 | 9 | 7 | 1 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 10 | 1 | 2 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 4 | 5 | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 5 | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT03729596/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03729596/SAP_001.pdf